CLINICAL TRIAL: NCT01425593
Title: T Cell Function in Chronic Idiopathic Urticaria
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0118-08-mmc; confino2009
Record Dates: First submitted 2011-08-28; First posted 2011-08-30 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-11

CONDITIONS: Chronic Urticaria
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — venous blood sample
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Chronic idiopathic urticaria (CIU) is a common form of chronic urticaria in which the cause is not detected after intensive clinical and laboratory investigation.In view of the current data, it was suggested that at least part of the patients with CIU have an autoimmune process.This study is designed to investigate the mechanisms involved in the regulation and activation of the immune cells in patients with CIU and corelate them with disease activity

ELIGIBILITY:
Inclusion Criteria:

* age above 18
* chronic urticaria

Exclusion Criteria:

* age below 18
* pregnancy
* other severe chronic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with chronic urticaria
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-03 (Actual); Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel